CLINICAL TRIAL: NCT05973838
Title: Peer-Delivered, Behavioral Activation Intervention to Improve Polysubstance Use and Retention in Mobile Telemedicine OUD Treatment in an Underserved, Rural Area
Brief Title: Peer Recovery to Improve Polysubstance Use and Mobile Telemedicine Retention
Acronym: PRISM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: University of Maryland, Baltimore (Other); Weill Medical College of Cornell University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jessica Magidson, Director and Associate Professor, University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1953327; R01DA057443 (NIH)
Record Dates: First submitted 2023-06-07; First posted 2023-08-03 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Polysubstance Addiction; Opioid Medication Assisted Treatment; Treatment Adherence; Retention in Care; Substance-Related Disorders
Keywords: Substance-Related Disorders; Opioid-Related Disorders; Polysubstance Use; Mental disorders
MeSH Terms: conditions — Treatment Adherence and Compliance; Substance-Related Disorders; Opioid-Related Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in parallel to receive either the Peer Activate intervention on the MTU or enhanced treatment as usual (TAU: treatment as usual services on the MTU in addition to referral to other available services in the community through study contact). Assessments will take place for both groups at baseline, at a midpoint (1-month), and follow ups at 3-month, 6-month and 12-months following the baseline assessment. Follow up assessments will be conducted by a blinded assessor.
Who Masked: Outcomes Assessor
Masking Description: At 3-month, 6-month and 12-months following the baseline assessment, a trained and randomization-blinded member of the research team will complete assessments with the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peer-Delivered Behavioral Activation ("Peer Activate") (Experimental): Participants in the Peer Activate intervention will receive a PRS-delivered behavioral activation intervention to address barriers to retention in methadone treatment and increase substance-free, positive reinforcement to support retention and reduce polysubstance use.
  Interventions: Behavioral: Peer-Delivered Behavioral Activation ("Peer Activate")
- Treatment As Usual (No Intervention): Participants in the TAU group will receive enhanced treatment as usual, defined as MTU services as usual enhanced with additional community referrals and follow-ups on those referrals, in addition to regular meetings with an addiction medicine physician and PRS on the MTU. Standard PRS contact typically includes connection to local resources and general peer support as needed.

INTERVENTIONS:
Behavioral: Peer-Delivered Behavioral Activation ("Peer Activate") — The PRS-delivered Peer Activate intervention will consist of approximately six weekly "core" sessions (approximately 30 minutes-1 hour), and then 6 optional "booster" sessions to reinforce skill practice. In Peer Activate sessions, participants will learn behavioral activation and problem-solving skills to reduce barriers to medication nonadherence and incorporate value-driven, substance-free, rewarding activities into their daily life to reduce polysubstance use and improve retention.
  Arms: Peer-Delivered Behavioral Activation ("Peer Activate")

SUMMARY:
The purpose of this study is to evaluate the feasibility and effectiveness of a peer-led, brief, behavioral intervention to improve adherence to medication for opioid use disorder (MOUD) and reduce polysubstance use among patients with OUD and polysubstance use in underserved areas. The intervention is based on behavioral activation (BA) and is specifically designed to be implemented by a trained peer recovery specialist. In this hybrid, Type-1 effectiveness-implementation randomized controlled trial (RCT), the investigators will evaluate the effectiveness and implementation of Peer Activate vs. treatment as usual (TAU) over twelve months.

DETAILED DESCRIPTION:
There is a significant burden of opioid and polysubstance use within the US. Yet many communities are poorly equipped to meet the pressing need for addiction treatment, including medications for OUD (MOUD) and evidence-based interventions (EBIs) to address the rise in opioid use disorder (OUD) and co-occurring stimulant use. The availability of telemedicine has helped fill the void of practitioners by providing buprenorphine for OUD treatment in underserved areas, however, OUD treatment retention remains an ongoing challenge, with polysubstance use and stimulant use exacerbating this. Peer recovery specialists (PRSs), trained individuals with their own lived experience with substance use disorder (SUD) and recovery, are a promising strategy to improve OUD treatment retention and polysubstance use at these sites using a reinforcement-based approach.

Behavioral activation (BA) may be a feasible, scalable, reinforcement-based approach for improving OUD treatment retention and reducing polysubstance use in underserved areas. By targeting increases in positive reinforcement, BA has been found to be effective for improving SUD treatment retention, preventing future relapse, including for stimulant use specifically, and improving medication adherence (i.e., for HIV) among low-income, minority populations with SUD as well as depression, which is a barrier to MOUD retention. BA has been shown to be feasibly delivered by peers and community health workers.

This study proposes to evaluate the effectiveness, implementation, and cost-effectiveness of an adapted PRS-delivered BA approach on the TM-MTU ("Peer Activate-MTU") compared to enhanced treatment as usual (ETAU; facilitated referrals and general PRS support) for patients with OUD and other polysubstance use receiving telemedicine buprenorphine. The investigators propose a randomized Type 1 hybrid effectiveness-implementation trial (n=180) to evaluate Peer Activate-MTU compared to ETAU. Specific aims are to evaluate the effectiveness of Peer Activate-MTU over 12-months on OUD treatment retention and polysubstance use. The investigators will also evaluate the implementation of Peer-Active-MTU, including feasibility, acceptability, fidelity, and adoption guided by RE-AIM.

ELIGIBILITY:
Inclusion Criteria:

Patient participants in the RCT must be 18 or older; receive OUD treatment as part of the telemedicine program; and exhibit polysubstance use within the past three-months (i.e., use of one or more non-prescribed substances (excluding opioids and/or tobacco) by urine toxicology or self-report.

Exclusion Criteria:

* Demonstrating active, unstable or untreated psychiatric symptoms, including mania and/or psychosis that would interfere with study participation
* Inability to understand the study and provide informed consent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Six-Month Polysubstance Use Urinalysis | Measured from baseline to 6-month follow-up
  Polysubstance use will be assessed using urinalysis. Urine samples are collected at each visit and sent out for toxicological analysis using a customized panel composed of 40 analytes, including both qualitative and quantitative results for opioids, stimulants, benzodiazepines, alcohol, marijuana, hallucinogens, methadone, buprenorphine and norbuprenorphine.
Six-Month Polysubstance Use Self Report | Assessed between the baseline assessment 6-month follow-up
  The New York University (NYU) polysubstance use measurement tool will be utilized to assess polysubstance frequency.

SECONDARY OUTCOMES:
Six-month OUD Treatment Retention | Measured from intake through 6-month follow up
  Retention is measured using chart review of clinic records of appointment attendance. Retention will be assessed measured as dichotomous retention (yes/no) at six months post MOUD initiation.
Six-month Buprenorphine Adherence | Measured from intake to six-month follow-up
  Buprenorphine adherence will be assessed through urinalysis. Urine samples are collected at each visit and sent out for toxicological analysis using a customized panel composed of 40 analytes, including both qualitative and quantitative results for opioids, stimulants, benzodiazepines, alcohol, marijuana, hallucinogens, methadone, buprenorphine and norbuprenorphine. Continuity of pharmacy for MOUD through 6 months will be assessed and calculated via the percent retained on MT for at least 6 months, defined as having one or more additional MOUD-related visits for each 30-day period up to 6 months.
Six-month Self-Report Buprenorphine Adherence | Assessed between the baseline assessment and 6-month follow-up
  The IRA Wilson will be utilized to assess self-report buprenorphine adherence
Six-Month Problems Associated with Substance Use | Assessed between the baseline assessment and 6-month follow-up
  Problems associated with use will be assessed using the Short Inventory of Problems (SIP), a 15-item measure that will be used to assess five domains of impairment related to polysubstance use.
Intervention Uptake | Assessed between the baseline assessment and 6-month follow-up
  Feasibility, defined as the suitability and practicability of the approach, will be measured quantitatively as the % of patients who agree to participate in the intervention.
Intervention Session Attendance | Assessed between the baseline assessment 6-month follow-up
  Acceptability, defined as satisfaction with or tolerability of the proposed approach, will be measured quantitatively by session attendance. Specifically, % of patients enrolled who attend ≥75% sessions will be measured.
Intervention Fidelity | Assessed at the acute post-treatment follow-up (approximately 3-months post-baseline assessment)
  Fidelity, defined as the delivery of the intervention as intended, will be measured based on PRS adherence to the intervention delivery. A random selection of 20% of sessions will be rated for fidelity by an independent rater, and % of intervention components delivered as intended will be measured.

OTHER OUTCOMES:
Three-month OUD Treatment Retention | Measured from intake through 3-month follow up
  Retention is measured using chart review of clinic records of appointment attendance. Retention will be assessed measured as dichotomous retention (yes/no) at three months post MOUD initiation.
Three-Month Polysubstance Use Urinalysis | Measured from baseline to 3-month follow-up.
  Polysubstance use will be assessed using urinalysis. Urine samples are collected at each visit and sent out for toxicological analysis using a customized panel composed of 40 analytes, including both qualitative and quantitative results for opioids, stimulants, benzodiazepines, alcohol, marijuana, hallucinogens, methadone, buprenorphine and norbuprenorphine.
Three-Month Polysubstance Use Self Report | Measured from baseline to 3-month follow-up.
  The New York University (NYU) polysubstance use measurement tool will be utilized to assess polysubstance frequency.
Three-Month Problems Associated with Substance Use | Assessed between baseline assessment and 3-month follow-up.
  Problems associated with use will be assessed using the Short Inventory of Problems (SIP), a 15-item measure that will be used to assess five domains of impairment related to polysubstance use.
Three-month Buprenorphine Adherence | Measured over 3 months
  Buprenorphine adherence will be assessed through urinalysis. Urine samples are collected at each visit and sent out for toxicological analysis using a customized panel composed of 40 analytes, including both qualitative and quantitative results for opioids, stimulants, benzodiazepines, alcohol, marijuana, hallucinogens, methadone, buprenorphine and norbuprenorphine. Continuity of pharmacy for MOUD through 3 months will be assessed and calculated via the percent retained on MT for at least 3 months, defined as having one or more additional MOUD-related visits for each 30-day period up to 3 months.
Three-month Self-Report Buprenorphine Adherence | Assessed between the baseline assessment and 3-month follow-up
  The IRA Wilson will be utilized to assess self-report buprenorphine adherence
Twelve-month OUD Treatment Retention | Measured from intake through 12-month follow up
  Retention is measured using chart review of clinic records of appointment attendance. Retention will be assessed measured as dichotomous retention (yes/no) at twelve months post MOUD initiation.
Twelve-Month Polysubstance Use Urinalysis | Measured from baseline to 12-month follow-up.
  Polysubstance use will be assessed using urinalysis. Urine samples are collected at each visit and sent out for toxicological analysis using a customized panel composed of 40 analytes, including both qualitative and quantitative results for opioids, stimulants, benzodiazepines, alcohol, marijuana, hallucinogens, methadone, buprenorphine and norbuprenorphine.
Twelve-Month Polysubstance Use Self Report | Measured from baseline to 12-month follow-up.
  The New York University (NYU) polysubstance use measurement tool will be utilized to assess polysubstance frequency.
Twelve-Month Problems Associated with Substance Use | Assessed between the baseline and 12-month follow-up.
  Problems associated with use will be assessed using the Short Inventory of Problems (SIP), a 15-item measure that will be used to assess five domains of impairment related to polysubstance use.
Twelve-month Buprenorphine Adherence | Measured over 12 months
  Buprenorphine adherence will be assessed through urinalysis. Urine samples are collected at each visit and sent out for toxicological analysis using a customized panel composed of 40 analytes, including both qualitative and quantitative results for opioids, stimulants, benzodiazepines, alcohol, marijuana, hallucinogens, methadone, buprenorphine and norbuprenorphine. Continuity of pharmacy for MOUD through 12 months will be assessed and calculated via the percent retained on MT for at least 12 months, defined as having one or more additional MOUD-related visits for each 30-day period up to 12 months.
Twelve-month Self-Report Buprenorphine Adherence | Assessed between the baseline assessment and 12-month follow-up
  The IRA Wilson will be utilized to assess self-report buprenorphine adherence
Six-month Treatment Cost | Measured from baseline to 6-month follow-up
  The resources required to implement and sustain the interventions (Peer Activate-MTU, and ETAU) will be identified via micro-costing techniques, using a tailored version of the Drug Abuse Treatment Cost Analysis Program (DATCAP) instrument, a standardized, customizable tool designed to capture intervention resources in multiple settings for the purpose of estimating costs.
Six-month Healthcare Resource Utilization | Measured from baseline to 6-month follow-up
  Healthcare Resource Utilization by participants will be self-reported using time-anchoring methodology via the Non-study Medical and Other Services (NMOS) form, and will include non-study MOUD care, inpatient, outpatient, and emergency department services; SUD treatment medications; residential and outpatient SUD treatment days; hospital SUD detoxification days; and mental health treatment.
Six-month Health-related Quality of Life | Measured from baseline to 6-month follow-up
  Health-related quality of life (HRQoL) will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS)-Preference (PROPr) instrument.
Six-month Non-Medical and Other Resource Utilization | Measured from baseline to 6-month follow-up
  Use of non-medical and other resources from the societal perspective (e.g., school/workplace productivity, travel time to care, caregiver burden, etc.) will also be self-reported using the NMOS.
Six-month Criminal and Legal Activities | Measured from baseline to 6-month follow-up
  Criminal and legal activities will be measured using the time-anchoring methodology via the Criminal-Legal Activities Form (CLAF).
Overdose risk | Measured from baseline to 6-month follow-up
  Overdose risk will be assessed as a binary outcome (including both fatal and non-fatal overdoses).

CONTACTS AND LOCATIONS:
Overall Officials: Jessica F Magidson, PhD, Principal Investigator — University of Maryland, College Park; Sarah M Kattakuzhy, MD, Principal Investigator — University of Maryland, Baltimore
Locations (4):
- United States (4):
  - HIPS Clinic, Washington D.C., District of Columbia
  - University of Maryland Baltimore (UMD Drug Treatment Center), Baltimore, Maryland
  - University of Maryland, College Park, College Park, Maryland
  - Caroline County Behavioral Health, Denton, Maryland

IPD SHARING:
Plan to Share IPD: Yes
After all primary analyses are complete, de-identified data will be uploaded to an NIH-supported data repository and/or available by request to the MPIs.

REFERENCES:
- [Background] Ghertner R. U.S. trends in the supply of providers with a waiver to prescribe buprenorphine for opioid use disorder in 2016 and 2018. Drug Alcohol Depend. 2019 Nov 1;204:107527. doi: 10.1016/j.drugalcdep.2019.06.029. Epub 2019 Aug 30. PMID 31525570
- [Background] Propst F, Rosenberg MP, Vande Woude GF. Proto-oncogene expression in germ cell development. Trends Genet. 1988 Jul;4(7):183-7. doi: 10.1016/0168-9525(88)90073-x. No abstract available. PMID 3070865
- [Background] McGeachie RE, Ford WJ, Nelson MJ, Elias D, Goldberg ME. Neuroradiology case of the day. AJR Am J Roentgenol. 1987 May;148(5):1053-7. doi: 10.2214/ajr.148.5.1053. No abstract available. PMID 3495110
- [Background] Reger KM, Hunter TB. Case of the month No. 67. Watch battery ingestion. Ariz Med. 1983 Aug;40(8):559-60. No abstract available. PMID 6625920
- [Background] Lees P, Allsup FC. Influence of oxytocin and growth hormone on the actions of aldosterone in the rat. Arch Int Pharmacodyn Ther. 1969 Feb;177(2):457-71. No abstract available. PMID 5807178
- [Background] Yamazaki F, Donaldson EM. Involvement of gonadotropin and steroid hormones in the spermiation of the goldfish (Carassius auratus). Gen Comp Endocrinol. 1969 Jun;12(3):491-7. doi: 10.1016/0016-6480(69)90165-8. No abstract available. PMID 4238929
- [Background] Koper S, Mucha M. A cineradiographic method for recording the function of the oesophageal groove in lambs. Acta Physiol Pol. 1983 Sep-Dec;34(5-6):539-45. PMID 6679990
- [Background] Delamothe T. Nursing grievances. I: Voting with their feet. Br Med J (Clin Res Ed). 1988 Jan 2;296(6614):25-8. doi: 10.1136/bmj.296.6614.25. No abstract available. PMID 3122920
- [Background] Tull MT, Berghoff CR, Bardeen JR, Schoenleber M, Konkle-Parker DJ. An Initial Open Trial of a Brief Behavioral Activation Treatment for Depression and Medication Adherence in HIV-Infected Patients. Behav Modif. 2018 Mar;42(2):196-209. doi: 10.1177/0145445517723901. Epub 2017 Aug 11. PMID 28799413
- [Background] Miyai K, Azukizawa M, Kumahara Y. Bioassay and immunoassay measurements of serum thyrotropin in primary hypothyroidism before and after the administration of thyrotropin releasing hormone. Horm Metab Res. 1974 Jan;6(1):9-12. doi: 10.1055/s-0028-1093894. No abstract available. PMID 4206586
- [Background] Kaye S. Insidious lead poisoning. Bol Asoc Med P R. 1967 Feb;59(2):63-70. No abstract available. PMID 4962865
- [Background] Richards DA, Ekers D, McMillan D, Taylor RS, Byford S, Warren FC, Barrett B, Farrand PA, Gilbody S, Kuyken W, O'Mahen H, Watkins ER, Wright KA, Hollon SD, Reed N, Rhodes S, Fletcher E, Finning K. Cost and Outcome of Behavioural Activation versus Cognitive Behavioural Therapy for Depression (COBRA): a randomised, controlled, non-inferiority trial. Lancet. 2016 Aug 27;388(10047):871-80. doi: 10.1016/S0140-6736(16)31140-0. Epub 2016 Jul 23. PMID 27461440
- [Background] VanderWilde RS, Pritchard DJ. Adamantinoma of the tibia. Orthopedics. 1992 Aug;15(8):950-3. doi: 10.3928/0147-7447-19920801-15. No abstract available. PMID 1508772
- [Background] Davison A, Tibbits G, Shi ZG, Moon J. Active oxygen in neuromuscular disorders. Mol Cell Biochem. 1988 Dec;84(2):199-216. doi: 10.1007/BF00421055. PMID 3068522
- [Background] Mack KA, Jones CM, Ballesteros MF. Illicit Drug Use, Illicit Drug Use Disorders, and Drug Overdose Deaths in Metropolitan and Nonmetropolitan Areas-United States. Am J Transplant. 2017 Dec;17(12):3241-3252. doi: 10.1111/ajt.14555. PMID 29145698
- [Background] Langabeer JR, Stotts AL, Cortez A, Tortolero G, Champagne-Langabeer T. Geographic proximity to buprenorphine treatment providers in the U.S. Drug Alcohol Depend. 2020 Aug 1;213:108131. doi: 10.1016/j.drugalcdep.2020.108131. Epub 2020 Jun 24. PMID 32599495
- [Background] Magidson JF, Kleinman MB, Bradley V, Anvari MS, Abidogun TM, Belcher AM, Greenblatt AD, Dean D, Hines A, Seitz-Brown CJ, Wagner M, Bennett M, Felton JW. Peer recovery specialist-delivered, behavioral activation intervention to improve retention in methadone treatment: Results from an open-label, Type 1 hybrid effectiveness-implementation pilot trial. Int J Drug Policy. 2022 Oct;108:103813. doi: 10.1016/j.drugpo.2022.103813. Epub 2022 Aug 3. PMID 35932644